CLINICAL TRIAL: NCT04912609
Title: An Observational Study in Subjects With Spastic Paraplegia Type 11 Taking Trehalose
Brief Title: Trehalose Administration in Subjects With Spastic Paraplegia 11 (3AL-SPG11)
Acronym: 3AL-SPG11
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Filippo Maria Santorelli, Director Molecular Medicine, Neurogenetics and Neuromuscular Disorders, IRCCS Fondazione Stella Maris
Other Study IDs: 3AL-SPG11
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Hereditary Spastic Paraplegia; Spastic Paraplegia Type 11
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Spastic paraplegia 11, autosomal recessive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hereditary spastic paraparesis type 11 (SPG11) is caused by mutations in the SPG11 gene that produces spatacsin, a protein involved in lysosomal function.

DETAILED DESCRIPTION:
Several experiments on subjects affected by neurodegenerative diseases with dysfunction of the autophagic-lysosomal system show that trehalose improves the pathological phenotype. This evidence indicates that trehalose could be used in patients with SPG11 to try to prevent the accumulation of glycosphingolipids at the lysosomal level and induce the genesis of new lysosomes. This study aims to record clinical data of 20 patients with SPG11 who take trehalose during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SPG11
* Written signed informed consent

Exclusion Criteria:

* Diagnosis of other concomitant neurodegenerative diseases
* taking other experimental drugs within 30 days of the first Study visit (T0) and during the study
* Refusal to sign informed consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be enrolled in our centre (IRCCS Fondazione Stella Maris) as part of the primary care during regular visits.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Spastic Paraplegia Rating Scale (SPRS) at 6 and 12 months | At baseline, month 6, month 12
  Assess changes in score of the Spastic Paraplegia Rating Scale (SPRS) over ± 10%

SECONDARY OUTCOMES:
Changes in glycosphingolipids and gangliosides plasmatic levels | At baseline, month 6, month 12
  Assess changes in glycosphingolipids and gangliosides plasmatic levels over ± 10%

CONTACTS AND LOCATIONS:
Overall Officials: Filippo M Santorelli, MD PhD, Principal Investigator — Filippo Santorelli-Lab Med Molecolare
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutry M, Branchu J, Lustremant C, Pujol C, Pernelle J, Matusiak R, Seyer A, Poirel M, Chu-Van E, Pierga A, Dobrenis K, Puech JP, Caillaud C, Durr A, Brice A, Colsch B, Mochel F, El Hachimi KH, Stevanin G, Darios F. Inhibition of Lysosome Membrane Recycling Causes Accumulation of Gangliosides that Contribute to Neurodegeneration. Cell Rep. 2018 Jun 26;23(13):3813-3826. doi: 10.1016/j.celrep.2018.05.098. PMID 29949766
- [Background] Branchu J, Boutry M, Sourd L, Depp M, Leone C, Corriger A, Vallucci M, Esteves T, Matusiak R, Dumont M, Muriel MP, Santorelli FM, Brice A, El Hachimi KH, Stevanin G, Darios F. Loss of spatacsin function alters lysosomal lipid clearance leading to upper and lower motor neuron degeneration. Neurobiol Dis. 2017 Jun;102:21-37. doi: 10.1016/j.nbd.2017.02.007. Epub 2017 Feb 22. PMID 28237315
- [Background] Chang J, Lee S, Blackstone C. Spastic paraplegia proteins spastizin and spatacsin mediate autophagic lysosome reformation. J Clin Invest. 2014 Dec;124(12):5249-62. doi: 10.1172/JCI77598. Epub 2014 Nov 3. PMID 25365221
- [Background] de Souza PVS, de Rezende Pinto WBV, de Rezende Batistella GN, Bortholin T, Oliveira ASB. Hereditary Spastic Paraplegia: Clinical and Genetic Hallmarks. Cerebellum. 2017 Apr;16(2):525-551. doi: 10.1007/s12311-016-0803-z. PMID 27271711
- [Background] Davies JE, Sarkar S, Rubinsztein DC. Trehalose reduces aggregate formation and delays pathology in a transgenic mouse model of oculopharyngeal muscular dystrophy. Hum Mol Genet. 2006 Jan 1;15(1):23-31. doi: 10.1093/hmg/ddi422. Epub 2005 Nov 25. PMID 16311254